CLINICAL TRIAL: NCT01905657
Title: A Phase II/III Randomized Trial of Two Doses of MK-3475 (SCH900475) Versus Docetaxel in Previously Treated Subjects With Non-Small Cell Lung Cancer
Brief Title: Study of Two Doses of Pembrolizumab (MK-3475) Versus Docetaxel in Previously Treated Participants With Non-Small Cell Lung Cancer (MK-3475-010/KEYNOTE-010)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-010; 2012-004391-19 (EudraCT Number); 132355 (Registry Identifier: Japic-CTI); MK-3475-010 (Other: Merck); KEYNOTE-010 (Other: Merck)
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Non Small Cell Lung Cancer (NSCLC)
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pembrolizumab 2 mg/kg (Experimental): Participants received pembrolizumab 2 mg/kg intravenously (IV) over 30 minutes Q3W for up to 2 years.
  Interventions: Biological: Pembrolizumab
- Pembrolizumab 10 mg/kg (Experimental): Participants received pembrolizumab 10 mg/kg IV over 30 minutes Q3W for up to 2 years.
  Interventions: Biological: Pembrolizumab
- Docetaxel 75 mg/m^2 (Active Comparator): Participants received docetaxel 75 mg/m^2 IV over 1 hour Q3W for up to 2 years.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab 10 mg/kg; Pembrolizumab 2 mg/kg
Drug: Docetaxel — IV infusion
  Other Names: TAXOTERE®
  Arms: Docetaxel 75 mg/m^2

SUMMARY:
This study compared two doses of pembrolizumab (MK-3475) versus docetaxel in participants with non-small cell lung cancer (NSCLC) who had experienced disease progression after platinum-containing systemic therapy. Participants were assigned randomly to receive either pembrolizumab 2 mg/kg once every three weeks (Q3W), pembrolizumab 10 mg/kg Q3W or docetaxel 75 mg/m^2 Q3W. The total number of participants randomized depended upon demonstration of sufficient objective responses at an interim analysis.

Eligible participants who were allocated to the first course of pembrolizumab (2 mg/kg Q3W or 10 mg/kg Q3W) and experienced disease progression, to be permitted to receive a second course of pembrolizumab as long as Inclusion/Exclusion criteria were met.

Protocol Amendment 12 (effective date: 09 Dec 2015) enabled eligible participants who were allocated to docetaxel and experienced disease progression, to be permitted to switch over to receive pembrolizumab 2 mg/kg Q3W as long as Inclusion/Exclusion criteria were met.

With Protocol Amendment 15 (effective date: 03 Jan 2018), all second course and switch over participants will receive pembrolizumab 200 mg Q3W. Response or progression during the second and switch over pembrolizumab courses will not count towards efficacy outcome measures, and adverse events during the second and switch over pembrolizumab courses will not count towards safety outcome measures.

Also with Amendment 15, once a participant has achieved the study objective or the study has ended, the participant will be discontinued from this study and enrolled in an extension study (Keynote 587; NCT03486873) to continue protocol-defined assessments and treatment. Switch over participants who have not transitioned to pembrolizumab will be considered for the extension study on a case-by-case basis.

The primary study hypotheses are that pembolizumab prolongs Overall Survival (OS) and Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by independent radiologists' review in previously-treated participants with NSCLC in the strongly positive programmed cell death ligand 1 (PD-L1) stratum compared to docetaxel and in participants whose tumors express PD-L1 compared to docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 3 months
* Histologically- or cytologically-confirmed diagnosis of NSCLC that is anti-programmed cell death ligand 1 (PD-L1) positive per central laboratory review
* At least one bi-dimensional measurable lesion
* Radiographic progression after treatment with at least 2 cycles of a platinum-containing doublet
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1

Exclusion Criteria:

* Prior therapy with docetaxel for NSCLC
* Receiving systemic steroid therapy within 3 days prior to the first dose of study treatment or receiving any other form of immunosuppressive medication
* Currently participating or has participated in a study using an investigational antineoplastic agent or device within 30 days of first dose
* Expected to require any other form of systemic or localized antineoplastic therapy while on trial
* History of allogeneic tissue/solid organ transplant
* Prior systemic cytotoxic chemotherapy, antineoplastic biological therapy (e.g., cetuximab), major surgery within 3 weeks of the first dose of study drug; received thoracic radiation therapy of >30 Gy within 6 months of the first dose of study drug; received prior tyrosine kinase inhibitor therapy or completed palliative radiotherapy within 7 days of the first dose of study drug
* Prior therapy with an anti-programmed cell death (PD)-1, anti-PD-L1, anti-PD-L2, anti-tumor necrosis factor CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways), or took part in another pembrolizumab trial
* Known history of prior malignancy, with the exception of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, or in situ cervical cancer, and has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Active autoimmune disease, or a documented history of autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents
* Interstitial lung disease, or history of pneumonitis requiring systemic steroids for treatment
* Known history or active human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial through 120 days after last dose of pembrolizumab or 180 days after last dose of docetaxel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1034 (Actual)
Dates: Start 2013-08-09 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Herbst RS, Baas P, Kim DW, Felip E, Perez-Gracia JL, Han JY, Molina J, Kim JH, Arvis CD, Ahn MJ, Majem M, Fidler MJ, de Castro G Jr, Garrido M, Lubiniecki GM, Shentu Y, Im E, Dolled-Filhart M, Garon EB. Pembrolizumab versus docetaxel for previously treated, PD-L1-positive, advanced non-small-cell lung cancer (KEYNOTE-010): a randomised controlled trial. Lancet. 2016 Apr 9;387(10027):1540-1550. doi: 10.1016/S0140-6736(15)01281-7. Epub 2015 Dec 19. PMID 26712084
- [Derived] Cristescu R, Aurora-Garg D, Albright A, Xu L, Liu XQ, Loboda A, Lang L, Jin F, Rubin EH, Snyder A, Lunceford J. Tumor mutational burden predicts the efficacy of pembrolizumab monotherapy: a pan-tumor retrospective analysis of participants with advanced solid tumors. J Immunother Cancer. 2022 Jan;10(1):e003091. doi: 10.1136/jitc-2021-003091. PMID 35101941
- [Derived] Jemielita T, Li XN, Piperdi B, Zhou W, Burke T, Chen C. Overall Survival With Second-Line Pembrolizumab in Patients With Non-Small-Cell Lung Cancer: Randomized Phase III Clinical Trial Versus Propensity-Adjusted Real-World Data. JCO Clin Cancer Inform. 2021 Jan;5:56-65. doi: 10.1200/CCI.20.00099. PMID 33439727
- [Derived] Lala M, Li TR, de Alwis DP, Sinha V, Mayawala K, Yamamoto N, Siu LL, Chartash E, Aboshady H, Jain L. A six-weekly dosing schedule for pembrolizumab in patients with cancer based on evaluation using modelling and simulation. Eur J Cancer. 2020 May;131:68-75. doi: 10.1016/j.ejca.2020.02.016. Epub 2020 Apr 15. PMID 32305010
- [Derived] Herbst RS, Garon EB, Kim DW, Cho BC, Perez-Gracia JL, Han JY, Arvis CD, Majem M, Forster MD, Monnet I, Novello S, Szalai Z, Gubens MA, Su WC, Ceresoli GL, Samkari A, Jensen EH, Lubiniecki GM, Baas P. Long-Term Outcomes and Retreatment Among Patients With Previously Treated, Programmed Death-Ligand 1-Positive, Advanced Non-Small-Cell Lung Cancer in the KEYNOTE-010 Study. J Clin Oncol. 2020 May 10;38(14):1580-1590. doi: 10.1200/JCO.19.02446. Epub 2020 Feb 20. PMID 32078391
- [Derived] van Vugt MJH, Stone JA, De Greef RHJMM, Snyder ES, Lipka L, Turner DC, Chain A, Lala M, Li M, Robey SH, Kondic AG, De Alwis D, Mayawala K, Jain L, Freshwater T. Immunogenicity of pembrolizumab in patients with advanced tumors. J Immunother Cancer. 2019 Aug 8;7(1):212. doi: 10.1186/s40425-019-0663-4. PMID 31395089
- [Derived] Barlesi F, Garon EB, Kim DW, Felip E, Han JY, Kim JH, Ahn MJ, Fidler MJ, Gubens MA, de Castro G Jr, Surmont V, Li Q, Deitz AC, Lubiniecki GM, Herbst RS. Health-Related Quality of Life in KEYNOTE-010: a Phase II/III Study of Pembrolizumab Versus Docetaxel in Patients With Previously Treated Advanced, Programmed Death Ligand 1-Expressing NSCLC. J Thorac Oncol. 2019 May;14(5):793-801. doi: 10.1016/j.jtho.2019.01.016. Epub 2019 Jan 31. PMID 30711649
- [Derived] Herbst RS, Baas P, Perez-Gracia JL, Felip E, Kim DW, Han JY, Molina JR, Kim JH, Dubos Arvis C, Ahn MJ, Majem M, Fidler MJ, Surmont V, de Castro G Jr, Garrido M, Shentu Y, Emancipator K, Samkari A, Jensen EH, Lubiniecki GM, Garon EB. Use of archival versus newly collected tumor samples for assessing PD-L1 expression and overall survival: an updated analysis of KEYNOTE-010 trial. Ann Oncol. 2019 Feb 1;30(2):281-289. doi: 10.1093/annonc/mdy545. PMID 30657853
- See also: Merck Oncology Clinical Trial Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had non-small cell lung cancer (NSCLC) and whose tumors were assessed as being programmed cell death ligand 1 (PD-L1) positive were recruited for this study.
Pre-assignment Details: Per protocol, response or progression during the second and switch over pembrolizumab courses was not counted towards efficacy outcome measures, and adverse events during the second and switch over pembrolizumab courses were not counted towards safety outcome measures.
  Final analyses for all primary and secondary outcome measures was done at the protocol-specified cutoff of 30-Sep-2015.
Groups:
- Pembrolizumab 2 mg/kg: Participants received pembrolizumab 2 mg/kg intravenously (IV) over 30 minutes every 3 weeks (Q3W) for up to 2 years. Qualified participants who received the first course of pembrolizumab 2 mg/kg Q3W for up to 2 years, but experienced disease progression, initiated a second course of pembrolizumab at the investigator's discretion, at 200 mg IV Q3W for up to 1 year.
- Pembrolizumab 10 mg/kg: Participants received pembrolizumab 10 mg/kg IV over 30 minutes Q3W for up to 2 years. Qualified participants who received the first course of pembrolizumab 10 mg/kg Q3W for up to 2 years, but experienced disease progression, initiated a second course of pembrolizumab at the investigator's discretion, at 200 mg IV Q3W for up to 1 year.
- Docetaxel 75 mg/m^2: Participants received docetaxel 75 mg/m^2 IV over 1 hour Q3W for up to 2 years. Qualified participants who received docetaxel 75 mg/m^2 Q3W for up to 2 years, but experienced disease progression, switched over to pembrolizumab, at the investigator's discretion, at 200 mg IV Q3W for up to 2 years.
Period: Overall Study
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Docetaxel 75 mg/m^2
Started | 345 | 346 | 343
Treated | 339 | 343 | 309
Received Second Course of Pembrolizumab | 14 | 7 | 0
Switched Over to Pembrolizumab | 0 | 0 | 8
Completed | 142 | 159 | 143
Not Completed | 203 | 187 | 200
Not completed — Adverse Event | 23 | 17 | 18
Not completed — Clinical Progression | 103 | 78 | 59
Not completed — Death | 40 | 43 | 47
Not completed — Excluded Medication | 13 | 16 | 9
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Physician Decision | 5 | 8 | 12
Not completed — Protocol Violation | 2 | 1 | 1
Not completed — Screen Failure | 0 | 1 | 0
Not completed — Withdrawal by Subject | 15 | 21 | 53
Not completed — Sponsor Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Docetaxel 75 mg/m^2 | Total
Number analyzed (Participants) | 345 | 346 | 343 | 1034
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.1 (9.6) | 62.3 (9.7) | 61.6 (9.8) | 62.0 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 133 | 134 | 399
  Male | 213 | 213 | 209 | 635
PD-L1 Tumor Expression Status [Count of Participants; unit: Participants] — PD-L1 expression was evaluated by immunohistochemistry (IHC) assay with a newly obtained tumor tissue with biopsy. If PD-L1 expression was observed in ≥1%, but ≤49% of tumor cells, a participant was categorized as weakly PD-L1 positive. If PD-L1 expression was observed in ≥50% of tumor cells, a participant was categorized as strongly PD-L1 positive.
  Participants
    Weakly PD-L1 Positive | 206 | 195 | 191 | 592
    Strongly PD-L1 Positive | 139 | 151 | 152 | 442

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. OS was analyzed using the Kaplan-Meier method and is reported in months. Per protocol, final analysis for this primary outcome measure was performed for the first pembrolizumab course and docetaxel treatment arms, with a protocol-specified analysis data cutoff date of 30 September (Sep) 2015.
Time Frame: Through pre-specified database cutoff date of 30 Sep 2015 (Up to approximately 24 months)
Population: Per protocol, OS for the first pembrolizumab course and docetaxel treatment arms was analyzed in all randomized participants who had strongly PD-L1 positive and all PD-L1 positive OS data available and usable. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Pembrolizumab 2 mg/kg: Participants received pembrolizumab 2 mg/kg IV over 30 minutes Q3W for up to 2 years. Qualified participants who received the first course of pembrolizumab 2 mg/kg Q3W for up to 2 years, but experienced disease progression, initiated a second course of pembrolizumab at the investigator's discretion, at 200 mg IV Q3W for up to 1 year.
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Docetaxel 75 mg/m^2
Number analyzed (Participants) | 344 | 346 | 343
Months
  Strongly PD-L1 Positive: number analyzed (Participants) | 139 | 151 | 152
  Strongly PD-L1 Positive | 14.9 [10.4 to NA] — Upper limit of OS not reached, due to insufficient number of deaths in the study. | 17.3 [11.8 to NA] — Upper limit of OS not reached, due to insufficient number of deaths in the study. | 8.2 [6.4 to 10.7]
  All PD-L1 Positive | 10.4 [9.4 to 11.9] | 12.7 [10.0 to 17.3] | 8.5 [7.5 to 9.8]
Statistical Analysis 1: Comparison: Pembrolizumab 2 mg/kg vs Docetaxel 75 mg/m^2; In participants with strongly PD-L1 positive tumors; Test type: Superiority or Other — Hazard Ratio based on stratified Cox regression model with treatment as a covariate and p-value based on stratified log-rank test, in accordance with the statistical analysis plan; p = 0.00024, Log Rank; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.38 to 0.77] — Numerator=Pembrolizumab 2 mg/kg Denominator=Docetaxel 75 mg/m^2
Statistical Analysis 2: Comparison: Pembrolizumab 10 mg/kg vs Docetaxel 75 mg/m^2; In participants with strongly PD-L1 positive tumors; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; p = 0.00002, Log Rank; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.36 to 0.70] — Numerator=Pembrolizumab 10 mg/kg Denominator=Docetaxel 75 mg/m^2
Statistical Analysis 3: Comparison: Pembrolizumab 2 mg/kg vs Docetaxel 75 mg/m^2; In participants with PD-L1 positive tumors; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; p = 0.00076, Log Rank; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.58 to 0.88] — Numerator=Pembrolizumab 2 mg/kg Denominator=Docetaxel 75 mg/m^2
Statistical Analysis 4: Comparison: Pembrolizumab 10 mg/kg vs Docetaxel 75 mg/m^2; In participants with PD-L1 positive tumors; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; p < 0.00001, Log Rank; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.49 to 0.75] — Numerator=Pembrolizumab 10 mg/kg Denominator=Docetaxel 75 mg/m^2

2. Primary Outcome: Progression-free Survival (PFS) by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS was defined as the time from the first day of study treatment to the first documented disease progression per RECIST 1.1 based on blinded independent central radiologists' review or death due to any cause, whichever occurred first. Using RECIST 1.1, progressive disease was defined as either a 20% relative increase in the sum of diameters of target lesions, taking as reference the smallest sum on study OR an absolute increase of >5 mm in the sum of lesions, OR the appearance of new lesions. PFS was analyzed using the Kaplan-Meier method and is reported in months. Per protocol, final analysis for this primary outcome measure was performed for the first pembrolizumab course and docetaxel treatment arms, with a protocol-specified analysis data cutoff date of 30 Sep 2015.
Time Frame: Through pre-specified database cutoff date of 30 Sep 2015 (Up to approximately 24 months)
Population: Per protocol, PFS for the first pembrolizumab course and docetaxel treatment arms was analyzed in all randomized participants who had strongly PD-L1 positive and all PD-L1 positive PFS data available and usable. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Docetaxel 75 mg/m^2
Number analyzed (Participants) | 344 | 346 | 343
Months
  Strongly PD-L1 Positive: number analyzed (Participants) | 139 | 151 | 152
  Strongly PD-L1 Positive | 5.2 [4.0 to 6.5] | 5.2 [4.1 to 8.1] | 4.1 [3.6 to 4.3]
  All PD-L1 Positive | 3.9 [3.1 to 4.1] | 4.0 [2.6 to 4.3] | 4.0 [3.1 to 4.2]
Statistical Analysis 1: Comparison: Pembrolizumab 2 mg/kg vs Docetaxel 75 mg/m^2; In participants with strongly PD-L1 positive tumors; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; p = 0.00009, Log Rank; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.43 to 0.77] — Numerator=Pembrolizumab 2 mg/kg Denominator=Docetaxel 75 mg/m^2
Statistical Analysis 2: Comparison: Pembrolizumab 10 mg/kg vs Docetaxel 75 mg/m^2; In participants with strongly PD-L1 positive tumors; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; p = 0.00007, Log Rank; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.45 to 0.78] — Numerator=Pembrolizumab 10 mg/kg Denominator=Docetaxel 75 mg/m^2
Statistical Analysis 3: Comparison: Pembrolizumab 2 mg/kg vs Docetaxel 75 mg/m^2; In participants with PD-L1 positive tumors; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; p = 0.06758, Log Rank; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.73 to 1.04] — Numerator=Pembrolizumab 2 mg/kg Denominator=Docetaxel 75 mg/m^2
Statistical Analysis 4: Comparison: Pembrolizumab 10 mg/kg vs Docetaxel 75 mg/m^2; In participants with PD-L1 positive tumors; Test type: Superiority or Other — [test comment as in outcome 1, analysis 1]; p = 0.00462, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.66 to 0.94] — Numerator=Pembrolizumab 10 mg/kg Denominator=Docetaxel 75 mg/m^2

3. Primary Outcome: Percentage of Participants Experiencing Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily had to have a causal relationship with this treatment. An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the study drug, was also an AE. Per protocol, final analysis for this primary outcome measure was performed for the first pembrolizumab course and docetaxel treatment arms, with a protocol-specified analysis data cutoff date of 30 Sep 2015.
Time Frame: Through pre-specified database cutoff date of 30 Sep 2015 (Up to approximately 24 months)
Population: Per protocol, participants experiencing AEs for the first pembrolizumab course and docetaxel treatment arms were analyzed in the All Participants As Treated (APAT) population. This consisted of all participants who received at least one dose of study drug. Participants were included in the treatment group based on the study treatment they received.
Measure: Number; unit: Percentage of Participants
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Docetaxel 75 mg/m^2
Number analyzed (Participants) | 339 | 343 | 309
Percentage of Participants | 97.6 | 96.2 | 96.1

4. Primary Outcome: Percentage of Participants Discontinuing Study Drug Due to AEs
Description: as for outcome 3
Time Frame: Through pre-specified database cutoff date of 30 Sep 2015 (Up to approximately 24 months)
Population: Per protocol, participants discontinuing study treatment due to AEs, for the first pembrolizumab course and docetaxel treatment arms were analyzed in the APAT population. This consisted of all participants who received at least one dose of study drug. Participants were included in the treatment group based on the study treatment they received.
Measure: Number; unit: Percentage of Participants
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Docetaxel 75 mg/m^2
Number analyzed (Participants) | 339 | 343 | 309
Percentage of Participants | 8.3 | 7.6 | 13.6

5. Secondary Outcome: Overall Response Rate (ORR) by RECIST 1.1
Description: ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR; disappearance of all target lesions) or Partial Response (PR; at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters) based on blinded independent central radiologists' review using RECIST 1.1. Per protocol, final analysis for this secondary outcome measure was performed for the first pembrolizumab course and docetaxel treatment arms, with a protocol-specified analysis data cutoff date of 30 Sep 2015.
Time Frame: Through pre-specified database cutoff date of 30 Sep 2015 (Up to approximately 24 months)
Population: Per protocol, ORR for the first pembrolizumab course and docetaxel treatment arms was analyzed in all randomized participants who had strongly PD-L1 positive and all PD-L1 positive ORR data available and usable. Participants were included in the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Docetaxel 75 mg/m^2
Number analyzed (Participants) | 344 | 346 | 343
Percentage of Participants
  Strongly PD-L1 Positive: number analyzed (Participants) | 139 | 151 | 152
  Strongly PD-L1 Positive | 30.2 [22.7 to 38.6] | 29.1 [22.0 to 37.1] | 7.9 [4.1 to 13.4]
  All PD-L1 Positive | 18.0 [14.1 to 22.5] | 18.5 [14.5 to 23.0] | 9.3 [6.5 to 12.9]
Statistical Analysis 1: Comparison: Pembrolizumab 2 mg/kg vs Pembrolizumab 10 mg/kg; In participants with strongly PD-L1 positive tumors; Test type: Superiority or Other; p = 0.66608, Miettinen & Nurminen method — P-value indicated for testing a difference in percentage equal to 0 versus a difference in percentage not equal to 0, in accordance with the statistical analysis plan; Difference in Percentages = -2.3, 95% CI 2-sided [-12.7 to 8.2] — This is an adjusted risk difference estimated by stratified Miettinen & Nurminen method
Statistical Analysis 2: Comparison: Pembrolizumab 10 mg/kg vs Docetaxel 75 mg/m^2; In participants with strongly PD-L1 positive tumors; Test type: Superiority or Other; p < 0.00001, Miettinen & Nurminen method — P-value indicated for testing a difference in percentage equal to 0 versus a difference in percentage greater than 0, in accordance with the statistical analysis plan; Difference in Percentages = 22.2, 95% CI 2-sided [14.0 to 30.7] — This is an adjusted risk difference estimated by stratified Miettinen & Nurminen method
Statistical Analysis 3: Comparison: Pembrolizumab 2 mg/kg vs Docetaxel 75 mg/m^2; In participants with PD-L1 positive tumors; Test type: Superiority or Other; p = 0.00045, Miettinen & Nurminen method — [p-value comment as in outcome 5, analysis 2]; Difference in Percentages = 8.7, 95% CI 2-sided [3.6 to 13.9] — This is an adjusted risk difference estimated by stratified Miettinen & Nurminen method
Statistical Analysis 4: Comparison: Pembrolizumab 10 mg/kg vs Docetaxel 75 mg/m^2; In participants with PD-L1 positive tumors; Test type: Superiority or Other; p = 0.00024, Miettinen & Nurminen method — [p-value comment as in outcome 5, analysis 2]; Difference in Percentages = 9.1, 95% CI 2-sided [4.1 to 14.3] — This is an adjusted risk difference estimated by stratified Miettinen & Nurminen method

6. Secondary Outcome: Duration of Response (DOR) by RECIST 1.1
Description: DOR is measured from the time measurement criteria were first met for CR/PR (whichever was first recorded) until the first date that death or progressive disease was objectively documented (taking as reference for progressive disease the smallest measurements recorded on study). Non-responders were not included in the analysis. DOR was analyzed using the Kaplan-Meier method and is reported in weeks. Per protocol, final analysis for this secondary outcome measure was performed for the first pembrolizumab course and docetaxel treatment arms, with a protocol-specified analysis data cutoff date of 30 Sep 2015.
Time Frame: Through pre-specified database cutoff date of 30 Sep 2015 (Up to approximately 24 months)
Population: Per protocol, DOR for the first pembrolizumab course and docetaxel treatment arms was analyzed in all randomized participants who demonstrated a CR/PR and had strongly PD-L1 positive and all PD-L1 positive DOR data available and usable. Participants were included in the treatment group to which they were randomized.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Docetaxel 75 mg/m^2
Number analyzed (Participants) | 62 | 64 | 32
Weeks
  Strongly PD-L1 Positive: number analyzed (Participants) | 42 | 44 | 12
  Strongly PD-L1 Positive | NA [3 to NA] — Median DOR and DOR upper limit not reached: No progressive disease by the time of last disease assessment. | NA [9 to NA] — Median DOR and DOR upper limit not reached: No progressive disease by the time of last disease assessment. | 35 [9 to NA] — DOR upper limit not reached: No progressive disease by the time of last disease assessment.
  All PD-L1 Positive | NA [3 to NA] — Median DOR and DOR upper limit not reached: No progressive disease by the time of last disease assessment. | NA [9 to NA] — Median DOR and DOR upper limit not reached: No progressive disease by the time of last disease assessment. | 27 [6 to NA] — DOR upper limit not reached: No progressive disease by the time of last disease assessment.

ADVERSE EVENTS:
Time Frame: Safety: Up to ~35 months for pembrolizumab first course and up to additional ~27 months for pembrolizumab second and switch over courses; All-cause mortality (ACM): Up to ~83 months for pembrolizumab first, second and switch over courses
Description: Safety and ACM were analyzed by treatment (pembrolizumab 2 mg/kg, 10 mg/kg, docetaxel 75 mg/m^2) and course (first, second, switch over). ACM was analyzed in all randomized participants and safety in all participants who got ≥1 dose of study drug. Per protocol disease progression of cancer was not considered an AE unless related to study drug. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression", "Disease progression" unrelated to study drug are excluded as AEs.
Groups:
- Pembrolizumab 2 mg/kg First Course: Participants received pembrolizumab 2 mg/kg IV over 30 minutes Q3W for up to 2 years.
- Pembrolizumab 10 mg/kg First Course: Participants received pembrolizumab 10 mg/kg IV over 30 minutes Q3W for up to 2 years.
- Pembrolizumab 2 mg/kg First Course to Pembrolizumab 200 mg Second Course: Qualified participants who received the first course of pembrolizumab 2 mg/kg Q3W for up to 2 years, but experienced disease progression, initiated a second course of pembrolizumab at the investigator's discretion, at 200 mg IV Q3W for up to 1 year.
- Pembrolizumab 10 mg/kg First Course to Pembrolizumab 200 mg Second Course: Qualified participants who received the first course of pembrolizumab 10 mg/kg Q3W for up to 2 years, but experienced disease progression, initiated a second course of pembrolizumab at the investigator's discretion, at 200 mg IV Q3W for up to 1 year.
- Docetaxel 75 mg/m^2 Switched Over to Pembrolizumab 200 mg: Qualified participants who received docetaxel 75 mg/m^2 Q3W for up to 2 years, but experienced disease progression, switched over to pembrolizumab, at the investigator's discretion, at 200 mg IV Q3W for up to 2 years.
Arm/Group | Pembrolizumab 2 mg/kg First Course | Pembrolizumab 10 mg/kg First Course | Docetaxel 75 mg/m^2 | Pembrolizumab 2 mg/kg First Course to Pembrolizumab 200 mg Second Course | Pembrolizumab 10 mg/kg First Course to Pembrolizumab 200 mg Second Course | Docetaxel 75 mg/m^2 Switched Over to Pembrolizumab 200 mg
All-Cause Mortality (participants affected / at risk) | 294/345 | 289/346 | 303/343 | 4/14 | 2/7 | 6/8
Serious Adverse Events (participants affected / at risk) | 124/339 | 133/343 | 107/309 | 5/14 | 2/7 | 1/8
Other Adverse Events (participants affected / at risk) | 312/339 | 301/343 | 279/309 | 9/14 | 5/7 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 2 mg/kg First Course (N=339) | Pembrolizumab 10 mg/kg First Course (N=343) | Docetaxel 75 mg/m^2 (N=309) | Pembrolizumab 2 mg/kg First Course to Pembrolizumab 200 mg Second Course (N=14) | Pembrolizumab 10 mg/kg First Course to Pembrolizumab 200 mg Second Course (N=7) | Docetaxel 75 mg/m^2 Switched Over to Pembrolizumab 200 mg (N=8)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 11 (11) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal suppression (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal hypomotility (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
External ear cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 20 (22) | 21 (22) | 19 (22) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyopneumothorax (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound sepsis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelitis transverse (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurological decompensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxic leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder hypertrophy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 6 (7) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 10 (10) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 8 (8) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary vascular disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infective spondylitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Pembrolizumab 2 mg/kg First Course (N=339) | Pembrolizumab 10 mg/kg First Course (N=343) | Docetaxel 75 mg/m^2 (N=309) | Pembrolizumab 2 mg/kg First Course to Pembrolizumab 200 mg Second Course (N=14) | Pembrolizumab 10 mg/kg First Course to Pembrolizumab 200 mg Second Course (N=7) | Docetaxel 75 mg/m^2 Switched Over to Pembrolizumab 200 mg (N=8)
Anaemia (Blood and lymphatic system disorders) | 37 (50) | 32 (43) | 61 (71) | 2 (3) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 47 (103) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 12 (13) | 19 (19) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 29 (30) | 29 (34) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 2 (2) | 2 (3) | 17 (18) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 20 (24) | 21 (23) | 13 (17) | 2 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 59 (65) | 57 (64) | 41 (47) | 1 (2) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 62 (91) | 51 (62) | 81 (111) | 1 (2) | 1 (1) | 2 (5)
Nausea (Gastrointestinal disorders) | 87 (105) | 75 (92) | 65 (80) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 19 (22) | 13 (15) | 49 (72) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 51 (60) | 48 (59) | 32 (37) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 44 (60) | 45 (59) | 51 (72) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 25 (26) | 32 (40) | 22 (23) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 102 (122) | 88 (107) | 106 (131) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 30 (35) | 28 (30) | 34 (37) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 51 (68) | 40 (64) | 42 (56) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 20 (26) | 23 (29) | 16 (16) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 18 (19) | 18 (26) | 11 (12) | 1 (2) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 19 (21) | 10 (12) | 9 (10) | 0 (0) | 1 (1) | 1 (5)
Alanine aminotransferase increased (Investigations) | 26 (35) | 20 (22) | 5 (6) | 1 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 20 (29) | 21 (24) | 4 (4) | 1 (2) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 12 (16) | 19 (19) | 5 (5) | 1 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 19 (26) | 17 (20) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (4) | 3 (4) | 25 (45) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 32 (37) | 33 (34) | 11 (13) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 3 (6) | 17 (29) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 104 (123) | 80 (93) | 74 (87) | 1 (1) | 2 (2) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 18 (27) | 15 (27) | 12 (13) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 48 (67) | 42 (50) | 29 (34) | 0 (0) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 41 (48) | 45 (51) | 23 (25) | 1 (2) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 39 (48) | 37 (41) | 10 (16) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 20 (28) | 15 (18) | 35 (52) | 0 (0) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 (23) | 26 (27) | 13 (16) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 30 (37) | 24 (26) | 12 (15) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 5 (5) | 8 (8) | 19 (24) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 42 (47) | 35 (43) | 22 (25) | 0 (0) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 8 (9) | 9 (9) | 37 (39) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 7 (9) | 8 (9) | 20 (22) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (7) | 6 (6) | 17 (17) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 18 (19) | 16 (16) | 9 (9) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 27 (29) | 22 (22) | 22 (24) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 82 (104) | 75 (94) | 43 (47) | 2 (2) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 81 (92) | 79 (95) | 65 (71) | 2 (2) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 26 (37) | 26 (33) | 20 (29) | 1 (1) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 21 (30) | 30 (32) | 10 (12) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (5) | 110 (112) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 15 (19) | 19 (25) | 8 (8) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 45 (62) | 52 (76) | 11 (11) | 4 (4) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 48 (62) | 59 (78) | 22 (22) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/6 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 6 (6) | 7 (7) | 0 (0) | 1 (1) | 0/6 (0)
Conjunctival haemorrhage (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 11 (11) | 12 (13) | 7 (7) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 10 (13) | 5 (6) | 14 (14) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (3) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 9 (15) | 12 (16) | 3 (6) | 1 (1) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 7 (9) | 3 (3) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 3 (5) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 8 (8) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraspinal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 14 (16) | 7 (12) | 9 (10) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 5 (6) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (5) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 5 (5) | 4 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 15 (20) | 5 (5) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Serum ferritin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6 (7) | 7 (8) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 10 (14) | 10 (15) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 15 (18) | 8 (16) | 11 (12) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 3 (3) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 4 (5) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 8 (8) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 8 (9) | 9 (9) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 12 (12) | 7 (7) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 7 (8) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (7) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 15 (16) | 12 (12) | 6 (7) | 0 (0) | 0 (0) | 1 (3)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT01905657/Prot_SAP_000.pdf